CLINICAL TRIAL: NCT04490057
Title: A Smart Approach to Treating Tobacco Use Disorder in Persons Living With HIV
Acronym: SMARTTT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2000026332; R01CA243910 (NIH)
Record Dates: First submitted 2020-07-22; First posted 2020-07-28 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum; Nicotine; Varenicline; Bupropion

STUDY DESIGN:
Intervention Model Description: Sequential multiple assignment randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- 12 wks NRT+CM / 12 wks NRT+CM (Experimental): Nicotine replacement therapy combined with contingency management. Responders remain on same treatment for second 12 weeks.
  Interventions: Drug: Nicotine patch, nicotine gum, nicotine nasal spray, nicotine inhaler; Behavioral: Contingency Management
- 12 wks NRT+CM/ 12 wks VAR or bupropion+CM (Experimental): Nicotine replacement therapy combined with contingency management. Non-responders switch to varenicline or bupropion combined with contingency management for second 12 weeks.
  Interventions: Drug: Nicotine patch, nicotine gum, nicotine nasal spray, nicotine inhaler; Drug: Varenicline or bupropion; Behavioral: Contingency Management
- 12 wks NRT+CM/12 wks NRT+CM plus (Experimental): Nicotine replacement therapy combined with contingency management Non-responders switch to nicotine replacement therapy combined with intensified contingency management for second 12 weeks.
  Interventions: Drug: Nicotine patch, nicotine gum, nicotine nasal spray, nicotine inhaler; Behavioral: Contingency Management
- 12 wks NRT/ 12 wks NRT (Experimental): Nicotine replacement therapy alone. Responders remain on nicotine replacement therapy.
  Interventions: Drug: Nicotine patch, nicotine gum, nicotine nasal spray, nicotine inhaler
- 12 wks NRT/ 12 wks VAR or bupropion (Experimental): Nicotine replacement therapy alone. Non-responders switch to varenicline or bupropion alone for second 12 weeks.
  Interventions: Drug: Nicotine patch, nicotine gum, nicotine nasal spray, nicotine inhaler; Drug: Varenicline or bupropion
- 12 wks NRT/ 12 wks NRT+CM (Experimental): Nicotine replacement therapy alone. Non-responders switch to nicotine replacement therapy combined with contingency management for second 12 weeks.
  Interventions: Drug: Nicotine patch, nicotine gum, nicotine nasal spray, nicotine inhaler; Behavioral: Contingency Management

INTERVENTIONS:
Drug: Nicotine patch, nicotine gum, nicotine nasal spray, nicotine inhaler — Participants will be prescribed both long-acting and short-acting nicotine replacement therapy.
Drug: Varenicline or bupropion — Participants will be prescribed varenicline (Chantix) or bupropion (Wellbutrin).
  Arms: 12 wks NRT+CM/ 12 wks VAR or bupropion+CM; 12 wks NRT/ 12 wks VAR or bupropion
Behavioral: Contingency Management — Participants will be financially rewarded for abstinence to tobacco.
  Arms: 12 wks NRT+CM / 12 wks NRT+CM; 12 wks NRT+CM/ 12 wks VAR or bupropion+CM; 12 wks NRT+CM/12 wks NRT+CM plus; 12 wks NRT/ 12 wks NRT+CM

SUMMARY:
Many people living with HIV (PLWH) smoke. Smoking in these individuals is often undertreated. This study plans to assess the ability of various clinical pathways involving tobacco treatment medications and contingency management (paying smokers for not smoking) to improve smoking cessation in a group of PLWH.

DETAILED DESCRIPTION:
Using a Sequential Multiple Assignment Randomized Trial (SMART) design, this project is a two-arm, two-stage randomized trial of 320 adult PWH who smoke cigarettes and receive care in one of three health systems (targeted enrollment changed from 632 to 320 with NCI approval and IRB protocol amendment). At inception, participants will be randomized to either combination nicotine replacement therapy (NRT, patch + short-acting NRT) or combination NRT+contingency management (CM). At 12 weeks, responders (non-smoking participants confirmed by exhaled carbon monoxide [eCO] or collateral verification) in both arms will receive 12 more weeks of the same treatment. Non-responders (participants with continued smoking by self-report and/or eCO) in both the NRT and NRT+CM arms will be re-randomized to 12 weeks of treatment, either with medication switch to oral medication, varenicline or bupropion, or intensified level of CM (start CM if no CM during first 12 weeks, or CM with higher reward schedule ["CM plus"] if NRT+CM group initially). The intervention will be delivered by trained clinical pharmacists. The primary outcomes will be self-reported reduction in average cigarettes smoked per day at 24 weeks and 12 weeks (primary outcome changed from eCO-confirmed abstinence to self-reported abstinence with NCI approval and IRB protocol amendment). The specific aims of the proposed study are to: (1) identify the optimal adaptive approach to promote reduced tobacco use (changed from eCO-confirmed smoking abstinence with NCI approval and protocol amendment) (2) study the effectiveness of various adaptive strategies on CD4 count, HIV viral suppression, and VACS index (validated measure of morbidity and mortality risk); and (3) grounded in implementation science and using aHybrid Effectiveness-Implementation Type I design, identify barriers and facilitators to delivering our intervention to inform future implementation.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive;
* >= 18 years old
* Receiving HIV care at Yale-New Haven Hospital, Bridgeport Hospital, Mount Sinai Hospital, or SUNY Downstate STAR clinic;
* Have smoked >= 100 cigarettes in lifetime;
* Currently smokes some days or every day;
* Smokes, on average, >= 5 cigarettes per day;
* Able to provide written informed consent.

Exclusion Criteria:

* Using only non-cigarette nicotine products (i.e., e-cigs, Juul, etc.);
* Currently using NRT, VAR, or bupropion (defined as use in the prior 7 days);
* Self-report or urine testing confirming pregnancy, nursing, or trying to conceive;
* Life-threatening or unstable medical, surgical, or psychiatric condition;
* Inability to provide at least one collateral contact (family member or friend);
* Living out of state;
* Unable to read or understand English (except at Mount Sinai site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Jennifer Edelman, MD, MHS, Principal Investigator — Yale University; Steven Bernstein, MD, Principal Investigator — Dartmouth College
Locations (4):
- United States (4):
  - Bridgeport Hospital Infectious Disease Clinic, Bridgeport, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut
  - SUNY Downstate STAR Clinic, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edelman EJ, Dziura J, Deng Y, Bold KW, Murphy SM, Porter E, Sigel KM, Yager JE, Ledgerwood DM, Bernstein SL. A SMARTTT approach to Treating Tobacco use disorder in persons with HIV (SMARTTT): Rationale and design for a hybrid type 1 effectiveness-implementation study. Contemp Clin Trials. 2021 Nov;110:106379. doi: 10.1016/j.cct.2021.106379. Epub 2021 Mar 29. PMID 33794354

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were consented, completed baseline and randomized to one of 2 arms in Stage 1: nicotine replacement therapy (NRT) or NRT+ CM (contingency management). At week 12, participants who were abstinent remained in their original arm. Participants who were not abstinent were re-randomized. If NRT in Stage 1, re-randomized to NRT+CM or varenicline (VAR). If NRT+CM Stage 1, re-randomized to NRT+CM intensified or VAR+CM.
Groups:
- Stage 1: NRT: Stage 1: participants randomized to receive nicotine replacement therapy only in Weeks 0-12
- Stage 1: NRT+CM: Participants randomized to receive nicotine replacement therapy and contingency management (Weeks 0-12)
- Stage 2: NRT Responders: Responders from Stage 1 remain on nicotine replacement therapy for Stage 2
- Stage 2: Varenicline or Bupropion: Non-responders to NRT in Stage 1 were switched to varenicline or bupropion alone for second 12 weeks (Stage 2).
- Stage 2: NRT+CM: Non-responders to NRT in Stage 1 were intensified to nicotine replacement therapy combined with contingency management for second 12 weeks (Stage 2).
- Stage 2: NRT+CM Responders: Responders to NRT+CM in Stage 1 remain on same treatment for second 12 weeks (Stage 2).
- Stage 2: Varenicline or Bupropion + CM: Non-responders NRT+CM in Stage 1 were switched to varenicline or bupropion combined with contingency management for second 12 weeks (Stage 2)
- Stage 2: NRT+CM Plus: Non-responders to NRT+CM in Stage 1 were switched to nicotine replacement therapy combined with intensified contingency management for second 12 weeks (Stage 2).
Period: Stage 1
Arm/Group | Stage 1: NRT | Stage 1: NRT+CM | Stage 2: NRT Responders | Stage 2: Varenicline or Bupropion | Stage 2: NRT+CM | Stage 2: NRT+CM Responders | Stage 2: Varenicline or Bupropion + CM | Stage 2: NRT+CM Plus
Started | 163 | 160 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 160 | 158 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Stage 2
Arm/Group | Stage 1: NRT | Stage 1: NRT+CM | Stage 2: NRT Responders | Stage 2: Varenicline or Bupropion | Stage 2: NRT+CM | Stage 2: NRT+CM Responders | Stage 2: Varenicline or Bupropion + CM | Stage 2: NRT+CM Plus
Started | 0 | 0 | 16 | 70 | 74 | 36 | 60 | 62
Completed | 0 | 0 | 16 | 59 | 56 | 32 | 39 | 48
Not Completed | 0 | 0 | 0 | 11 | 18 | 4 | 21 | 14
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 11 | 17 | 4 | 21 | 14

BASELINE CHARACTERISTICS:
Population: Includes all participants who started Stage 1
Groups:
- Stage 1: Nicotine Replacement Only (NRT): Participants met with a clinical pharmacist 6 times (baseline visit plus 5 follow-up visits) for nicotine replacement therapy prescriptions and tobacco cessation counseling
- Stage 1: Nicotine Replacement (NRT) + Contingency Management (CM): Participants met with a clinical pharmacist 6 times (baseline visit plus 5 follow-up visits) for nicotine replacement (NRT) prescriptions and tobacco cessation counseling. Participants in the NRT+CM arm also had the opportunity to earn prizes (gift cards) for tobacco abstinence, verified by exhaled carbon monoxide or next closest informant verification.
- Total: Total of all reporting groups
Arm/Group | Stage 1: Nicotine Replacement Only (NRT) | Stage 1: Nicotine Replacement (NRT) + Contingency Management (CM) | Total
Number analyzed (Participants) | 163 | 160 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years
  years | 55.71 (10.8) | 54.42 (10.6) | 55.08 (10.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 71 | 142
  Male | 92 | 89 | 181
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 3 | 8
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 116 | 114 | 230
  White | 29 | 33 | 62
  More than one race | 9 | 6 | 15
  Unknown or Not Reported | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 42 | 74
  Not Hispanic or Latino | 130 | 118 | 248
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: Participants]
  United States | 163 | 160 | 323
Cigarettes per day [Median (Inter-Quartile Range); unit: cigarettes per day] — Number of cigarettes smoked per day
  cigarettes per day | 10.0 [8.0 to 20.0] | 10.0 [7.0 to 17.5] | 10.0 [7.0 to 20.0]
Exhaled carbon monoxide at baseline [Median (Inter-Quartile Range); unit: parts per million (ppm)] — exhaled carbon monoxide at baseline, measured in parts per million (ppm) Population: eCO was not collected for 5 participants at baseline due to staff error.
  parts per million (ppm)
    number analyzed (Participants) | 159 | 159 | 318
    (all) | 10.0 [6.0 to 16.0] | 10.0 [6.0 to 16.0] | 10.0 [6.0 to 16.0]
VACS 2.0 score [Median (Inter-Quartile Range); unit: score on a scale] — The Veterans Aging Cohort Study (VACS) 2.0 Index is A validated measure of morbidity and mortality. It estimates risk of 5-year all-cause mortality in patients with HIV. Total score range of 0-129. A higher total score indicates a greater risk of adverse health outcomes. Population: 8 participants were missing a lab value required to calculate VACS 2.0
  score on a scale
    number analyzed (Participants) | 159 | 156 | 315
    (all) | 45.0 [31.0 to 58.0] | 42.0 [33.0 to 53.0] | 43.0 [32.0 to 56.0]
HIV viral load, detectable [Count of Participants; unit: Participants] — HIV viral load greater than 200 copies per milliliter of blood and detectable on standard lab test Population: HIV viral load was not available at baseline for 3 participants
  Participants
    number analyzed (Participants) | 162 | 158 | 320
    Viral load detectable | 19 | 17 | 36
    Viral load not detectable | 143 | 141 | 284
CD4 cell count [Median (Inter-Quartile Range); unit: cells per cubic millimeter] — CD4 lymphocyte cell count. Normal range is 500-1200 cells per cubic millimeter. As HIV infection progresses, CD4 count drops. Population: CD4 count was not available for 1 participant at baseline
  cells per cubic millimeter
    number analyzed (Participants) | 162 | 160 | 322
    (all) | 600.0 [331.0 to 875.0] | 596.5 [356.0 to 867.5] | 596.5 [352.0 to 875.0]

OUTCOME MEASURES:

1. Primary Outcome: Self Reported Reduction in Average Cigarettes Smoked Per Day at 12 Weeks
Description: Self reported reduction in average cigarettes smoked per day at 12 weeks
Time Frame: Week 12
Measure: Least Squares Mean (97.5% Confidence Interval); unit: cigarettes per day
Arm/Group | Stage 1: Nicotine Replacement only (NRT) | Stage 1: Nicotine Replacement (NRT) + Contingency Management (CM)
Number analyzed (Participants) | 163 | 160
cigarettes per day | 5.2 [3.9 to 6.5] | 4.9 [3.5 to 6.2]

2. Primary Outcome: Self Reported Reduction in Average Cigarettes Smoked Per Day at 24 Weeks
Description: Self reported reduction in cigarettes smoked per day at 24 weeks
Time Frame: 24 weeks
Measure: Least Squares Mean (99% Confidence Interval); unit: cigarettes per day
Arm/Group | Stage 2: NRT responders | Stage 2: varenicline or bupropion | Stage 2: NRT+CM | Stage 2: NRT+CM responders | Stage 2: varenicline or bupropion + CM | Stage 2: NRT+CM plus
Number analyzed (Participants) | 16 | 59 | 56 | 32 | 39 | 48
cigarettes per day | 7.90 [4.355 to 11.44] | 6.23 [4.45 to 8.02] | 2.97 [1.50 to 4.44] | 10.92 [8.40 to 13.43] | 4.00 [2.48 to 5.52] | 4.20 [2.60 to 5.80]

3. Secondary Outcome: Exhaled Carbon Monoxide (eCO) Confirmed Smoking Abstinence at 12 Weeks
Description: Number of participants with smoking abstinence confirmed by exhaled carbon monoxide or next closest informant verification
Time Frame: 12 weeks from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 1: Nicotine Replacement only (NRT) | Stage 1: Nicotine Replacement (NRT) + Contingency Management (CM)
Number analyzed (Participants) | 163 | 160
Participants | 16 [3.3 to 18.7] | 36 [9.8 to 36.8]

4. Secondary Outcome: Exhaled Carbon Monoxide (eCO) Confirmed Smoking Abstinence at 24 Weeks
Description: as for outcome 3
Time Frame: 24 weeks from baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: NRT responders | Stage 2: varenicline or bupropion | Stage 2: NRT+CM | Stage 2: NRT+CM responders | Stage 2: varenicline or bupropion + CM | Stage 2: NRT+CM plus
Number analyzed (Participants) | 16 | 59 | 56 | 32 | 39 | 48
Participants | 4 [4.55 to 59.91] | 6 [4.58 to 32.82] | 7 [6.43 to 32.21] | 23 [47.77 to 89.36] | 3 [11.58 to 48.44] | 8 [15.61 to 53.04]

5. Secondary Outcome: VACS Index 2.0 Score
Description: The Veterans Aging Cohort Study (VACS) 2.0 Index is A validated measure of morbidity and mortality. It estimates risk of 5-year all-cause mortality in patients with HIV. Total score range of 0-129. A higher total score indicates a greater risk of adverse health outcomes.
Time Frame: 24 weeks from baseline
Population: Lab results were collected for all participants at Week 24 including those who did not complete the Week 24 assessment battery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Stage 2: NRT responders | Stage 2: varenicline or bupropion | Stage 2: NRT+CM | Stage 2: NRT+CM responders | Stage 2: varenicline or bupropion + CM | Stage 2: NRT+CM plus
Number analyzed (Participants) | 16 | 70 | 69 | 34 | 59 | 60
score on a scale | 42.88 (15.09) | 47.26 (17.61) | 49.42 (19.61) | 42.65 (15.38) | 42.66 (15.66) | 43.63 (15.70)

6. Secondary Outcome: CD4 Count
Description: CD4 lymphocyte cell count. Normal range is 500-1200 cells per cubic millimeter. As HIV infection progresses, CD4 count drops.
Time Frame: 24 weeks from baseline
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Cells per cubic millimeter
Arm/Group | Stage 2: NRT responders | Stage 2: varenicline or bupropion | Stage 2: NRT+CM | Stage 2: NRT+CM responders | Stage 2: varenicline or bupropion + CM | Stage 2: NRT+CM plus
Number analyzed (Participants) | 16 | 70 | 69 | 35 | 59 | 60
Cells per cubic millimeter | 668.00 (384.08) | 576.53 (347.76) | 648.38 (423.08) | 640.57 (370.12) | 724.92 (521.86) | 696.97 (421.36)

7. Secondary Outcome: HIV Viral Load, Detectable
Description: HIV viral load greater than 200 copies per milliliter of blood and detectable on standard lab test
Time Frame: 24 weeks from baseline
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Stage 2: NRT responders | Stage 2: varenicline or bupropion | Stage 2: NRT+CM | Stage 2: NRT+CM responders | Stage 2: varenicline or bupropion + CM | Stage 2: NRT+CM plus
Number analyzed (Participants) | 15 | 70 | 74 | 34 | 60 | 62
Participants | 0 | 10 | 14 | 3 | 5 | 7

ADVERSE EVENTS:
Time Frame: Stage 1: up to 12 weeks; Stage 2: up to 24 weeks
Arm/Group | Stage 1: NRT | Stage 1: NRT+CM | Stage 2: NRT Responders | Stage 2: Varenicline or Bupropion | Stage 2: NRT+CM | Stage 2: NRT+CM Responders | Stage 2: Varenicline or Bupropion + CM | Stage 2: NRT+CM Plus
All-Cause Mortality (participants affected / at risk) | 1/163 | 2/160 | 0/16 | 0/70 | 1/74 | 0/36 | 0/60 | 0/62
Serious Adverse Events (participants affected / at risk) | 13/163 | 9/160 | 1/16 | 5/70 | 4/74 | 1/36 | 3/60 | 3/62
Other Adverse Events (participants affected / at risk) | 6/163 | 14/160 | 0/16 | 2/70 | 0/74 | 1/36 | 3/60 | 2/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: NRT (N=163) | Stage 1: NRT+CM (N=160) | Stage 2: NRT Responders (N=16) | Stage 2: Varenicline or Bupropion (N=70) | Stage 2: NRT+CM (N=74) | Stage 2: NRT+CM Responders (N=36) | Stage 2: Varenicline or Bupropion + CM (N=60) | Stage 2: NRT+CM Plus (N=62)
Gastrointestinal (nausea, diarrhea, abdominal pain) (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection - pathogen unspecified (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint pain or connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver injury or dysfunction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurological disorders (sedation, lethargy, dizziness) (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorders including pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Altered mental status (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol withdrawal (Social circumstances) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Other (Social circumstances) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidality (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac illness or injury (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1: NRT (N=163) | Stage 1: NRT+CM (N=160) | Stage 2: NRT Responders (N=16) | Stage 2: Varenicline or Bupropion (N=70) | Stage 2: NRT+CM (N=74) | Stage 2: NRT+CM Responders (N=36) | Stage 2: Varenicline or Bupropion + CM (N=60) | Stage 2: NRT+CM Plus (N=62)
Gastrointestinal Gastrointestinal (nausea, diarrhea, abdominal pain) (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac illness or injury (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver injury or dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorders including pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Reaction to nicotine replacement therapy (Product Issues) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Anticipated side effects of nicotine replacement therapy: sleep disturbances, jittery/shaking, etc.
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Psychiatric issues (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
1. The COVID-19 pandemic delayed enrollment leading to a reduction in sample size and change in endpoint to reduction in # of cigarettes/day. Due to these changes, we may have been underpowered to detect improved abstinence in Stage 2. 2. Participants were given prescriptions for medication, not actual medication and we observed access issues. 3. The study was conducted in urban HIV clinics in the Northeast US which may limit generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT04490057/Prot_SAP_001.pdf
  • Informed Consent Form (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT04490057/ICF_002.pdf